CLINICAL TRIAL: NCT01091740
Title: ComparisiOn of Neointimal coVerage betwEen zotaRolimus Eluting Stent and Everolimus Eluting Stent Using Optical Coherence Tomography at 3 Months
Brief Title: ComparisiOn of Neointimal coVerage betwEen ZES and EES Using OCT at 3 Months
Acronym: COVER OCT-II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jung-Sun Kim, Assistant Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2009-0010
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Artery Disease
Keywords: Drug eluting stent; Tomography, optical coherence
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZES resolute (Endeavor Resolute) (Experimental)
  Interventions: Device: ZES resolute (Endeavor Resolute)
- EES (Xience) (Active Comparator)
  Interventions: Device: EES (Xience)

INTERVENTIONS:
Device: ZES resolute (Endeavor Resolute) — 2nd generation drug eluting stent, which is coated with zotarolimus
  Other Names: Endeavor resolute
  Arms: ZES resolute (Endeavor Resolute)
Device: EES (Xience) — 2nd generation drug eluting stent, which is coated with everolimus
  Other Names: Xience
  Arms: EES (Xience)

SUMMARY:
This study try to 1) evaluate the neointimal coverage and malapposition at 3 month after new zotarolimus eluting stent (Endeavor resolute) and everolimus eluting stent (Xience) implantation and 2) compare them between ZES resolute and EES at 3 months (early period) after stent implantation.

DETAILED DESCRIPTION:
Recent autopsy study showed the most important histological and morphometric predictors of stent thrombosis were endothelial coverage and the ratio of uncovered to total strut after drug eluting stent (DES) implantation. Although there have been some controversies, incomplete stent apposition might be possible cause of very late stent thrombosis after DES implantation. Therefore, theoretically dual antiplatelet therapy should be continued to prevent the stent thrombosis until complete reendothelialization. But, detection of endothelial coverage over stent is not possible with available intravascular devices in clinical practice. Among currently available intravascular devices, intravascular optical coherence tomography (OCT) could give a more clear identification for a thin layer of neointimal hyperplasia (NIH) and malapposition with high-resolution (10 -20 μm) compared to intravascular ultrasound (100-150 μm). Previous OCT studies showed the significant different pattern of neointimal coverage between baremetal stent (BMS) and DES. In our experience, there were also some differences in neointimal coverage among the DESs, especially in zotarolimus eluting stent (ZES). ZES have been known to be associated with significantly more neointimal coverage than SES at 8 months intravascular untrasound (IVUS). This finding might be related with strut thickness and drug elution property. In our data, 99.7 % of stent struts were covered with neointima in ZES, but 93.2 % in sirolimus eluting stent (SES) at 9 month follow-up OCT. This difference was more distinct in patients with acute myocardial infarction (99.3 % in ZES vs.79.9 % in SES).

Both everolimus eluting stent (EES) was recently introduced and ZES resolute also will be available in the near future in Korea. Previous phosphorylcholine polymer was replaced with new, proprietary polymer which can provide extended elution kinetics in ZES resolute. Therefore, efficacy to suppress the neointimal growth might be improved but, safety for neointimal coverage needs to be evaluated in human coronary artery. Both new DESs are cobalt chrominum stent with thin stent strut and reported similar efficacy for suppressing the neointima growth. Also, endothelial coverage over stent strut occurred earlier compared to previous DESs (SES or PES) in animal experiments. But, there has been no data for neointimal coverage and malapposition of ZES resolute and EES using OCT in human coronary artery.

Recent paper according to Kubo et al reported that serial OCT examinations demonstrated markedly different vascular response up to 9 months after SES implantation between unstable angina and stable angina patients. These findings implied that initial native vessel status, which covered with stent, might be important and related with neoinitmal coverage and malapposition. But, there is little data evaluated the relationship between initial lesion status and neointimal coverage or late malapposition with OCT.

Therefore, this study will 1) evaluate the neointimal coverage and malapposition at 3 month after ZES resolute and EES implantation and 2) compare them between ZES resolute and EES at 3 months after stent implantation.

2. STUDY OBJECTIVE This study is an prospective open labeled randomized study to compare the neointimal coverage of ZES resolute (Endeavor® resolute) and EES (Xience®) in 3 month after stent implantation by OCT.

2.1. Primary end point The primary endpoint is to compare the pattern of neointimal coverage between ZES resoute (Endeavor® resolute) and EES (Xience®) at 3 months after stent implantation by OCT.

2.2. Secondary end point The secondary objective of this study is to evaluate neointimal growth between ZES resolute and EES at 3 months and 2) to compare the difference in early and late malapposition between ZES resolute and EES at 3 months.

3. Methods and Design

3.1 Patient enrollment Patients with stable angina pectoris who present to the cath lab for non-emergent PCI are eligible for participation. A patient is considered to be enrolled if they meet all of the inclusion and have none of the exclusion criteria.

Inclusion criteria

* Significant coronary de novo lesion (> 70% by quantitative angiographic analysis)
* Patients with stable angina pectoris who are considered for coronary revascularization.
* Reference vessel diameter of 2.5 to 3.5 mm by operator assessment

Exclusion criteria

The criteria for exclusion were

* Acute coronary syndrome
* Contraindication to anti-platelet agents
* Proximal leison within 15 mm from ostium
* Treated with any DES within 1 year at other vessel
* Creatinine level 2.0 mg/dL or ESRD
* Severe hepatic dysfunction (3 times normal reference values)
* Pregnant women or women with potential childbearing
* Complex lesion morphologies (aorto-ostial, unprotected Left main, chronic total occlusion)
* Target lesion is vein graft lesion
* Reference vessel < 2.5 mm or > 4.0mm diameter by visual

3.2. Sample Size and Statistical analysis

Calculation of the sample size could not be done because of observation study. Therefore, we decided to enroll 40 patients for 20 ZESs resolute and 20 EESs considering sufficient stent strut (over 3000 stent struts each group).

Results are expressed as the mean ±SD. Comparisons of discrete variables were made using the chi-square test or Fisher's Exact Test. Student t-tests were used for continuous variables. Because the distribution was skewed due to a small study sample, non-parametric tests (Mann-Whitney test for unpaired variables and Wilcoxon-signed rank test for paired variables) were used. All statistical analysis was performed with SPSS 13.0. (SPSS Inc., Chicago, IL, USA). A value of p<0.05 was considered statistically significant.

4. STUDY PROCEDURE

The cath lab will follow site standard operating procedures for PTCA and stenting. Stent overlapping is not allowed. Treatment of multiple vessels is acceptable. However, information will be collected on only one study lesion per patient.

Information will be collected and recorded on the treated study vessel including angiographic, IVUS and OCT parameters. The IVUS and OCT study should be checked in the procedure and follow up at 3 months angiography.

4.1. PROCEDURAL MATERIALS Endeavor ® resolute 2.75 to 3.5 mm All available length Drug Eluting Stent Xience ® 2.75 to 3.5 mm All available length

4.2 RANDOMIZATION Patients with native coronary arteries who fulfill all enrollment criteria will be randomized to receive either ZES (Endeavor®) resolute or EES (Xience or Promus®). Randomization will be performed in a 1:1 ratio of ZES or EES according to each clinical presentation.

4.3 STENT SELECTION The vessel size will be determined either by quantitative angiography or by IVUS for appropriate stent size selection.

4.4 IVUS ASSESSMENT IVUS assessment was performed using a commercially available IVUS system (Boston Scientific/ Scimed, Natick, MA). Studies were recorded on Index system (Echoplaque 2; INDEC Systems Inc, Mountain View, CA) for off-line analysis. Motorized transducer pullback permitted cross-sectional area measurements at 1mm axial increments throughout the length of the stent. All IVUS studies were performed after the intracoronary administration of 200 µg of nitroglycerin. The reference segment was the most visually normal cross section (largest lumen with least plaque burden) within 10mm proximal or distal to the lesion. Using the software, external elastic membrane (EEM) CSA (mm2), lumen CSA (mm2), minimal stent cross-sectional area (MSA); identified as the CSA at the tightest segment within stent, stent MLD were determined. The CSA at the proximal and the distal reference segments and at the most stenotic lesion as well as the CSA at the proximal and the distal stent edge was determined. A determination of the percent expansion was made by measuring the MSA and the average reference segment CSA. Average reference segment CSA is calculated as [Proximal Reference segment CSA +Distal Reference segment CSA)/2]. Plaque volume was calculated as vessel minus stent volume. Neointimal volume was calculated as stent minus lumen volume, and percentage (%) of neointimal obstruction was calculated as neointimal volume divided by stent volume. Neointimal coverage over stent surface and mean physical neointimal thickness were obtained by measuring circumferential stent length covered with neointimal hyperplasia (LN) and stent perimeter (LS) at every 1-mm cross-sectional image throughout the stented segment: (a) percentage of neointimal coverage over stent surface, calculated as total LN divided by total LS, and (b) mean physical neointimal thickness, calculated as mean neointimal area divided by mean LN for only the cross sections with detectable neointima.

4.5. OCT ASSESSMENT OCT measurements will be made as following methods: (Takano M, et al. Evaluation by Optical Coherence Tomography of Neointimal Coverage of Sirolimus-Eluting Stent Three Months After Implantation. Am J Cardiol 2007;99: 10331038)

Cross-sectional OCT images were analyzed at 1-mm intervals (every 15 frames). Neointimal hyperplasia (NIH) thickness inside stent struts was measured. Stent area and lumen area in every image were measured by manual trace and percent NIH area was calculated as percent NIH area = ([stent area - lumen area]/ stent area) / 100. Measured NIH thickness equal to 0 micro meter was defined as exposure, and maximum distance > 110 micro meter between the strut surface and adjacent vessel surface (thickness of strut and polymer) was defined as malapposition. On an image of stent malapposition, lumen area was divided into an in-stent lumen area and an extra-stent lumen area. . Intracoronary thrombus was defined as a protruding mass beyond the stent strut into the lumen. Bifurcation lesions with major sidebranches were excluded from this analysis. Inter- and intraobserver variabilities were assessed by evaluation of 20 random cross- sectional images by 2 independent readers and by the same reader at 2 separate time points, respectively.

4.6. Follow-Up

All patients will be followed after hospital discharge. When patients come back in 3 and 9 months after the discharge due to clinical follow-up, the patient record will be updated.

1. Clinical follow-up at 3, 9 months and 2 years after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Significant coronary de novo lesion (> 70% by quantitative angiographic analysis)
* Patients with stable angina pectoris who are considered for coronary revascularization.
* Reference vessel diameter of 2.5 to 3.5 mm by operator assessment

Exclusion Criteria:

* Acute coronary syndrome
* Contraindication to anti-platelet agents
* Proximal leison within 15 mm from ostium
* Treated with any DES within 1 year at other vessel
* Creatinine level 2.0 mg/dL or ESRD
* Severe hepatic dysfunction (3 times normal reference values)
* Pregnant women or women with potential childbearing
* Complex lesion morphologies (aorto-ostial, unprotected Left main, chronic total occlusion)
* Target lesion is vein graft lesion
* Reference vessel < 2.5 mm or > 4.0mm diameter by visual

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The rate of neointimal coverage between ZES resolute and EES at 3 months after stent implantation by OCT. | 3 months after stent implantation

SECONDARY OUTCOMES:
Neointimal growth between ZES resolute and EES at 3 months after stent by OCT. | 3 months after stent implantation
Early malapposition just after stent implantation and late malapposition at 3 months after stent implantaiton between ZES resolute and EES by OCT. | 3 months after stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Sun Kim, MD, Ph D, Principal Investigator — Division of Cardiology, Cardiovascular Hospital, Yonsei University
Locations (2):
- South Korea (2):
  - Dongsan Medical Center, Keimyung University College of Medicine, Daegu
  - Division of Cardiology, Cardiovascular Hospital, Yonsei University, Seoul